CLINICAL TRIAL: NCT06994208
Title: Demographic, Clinical, Dermoscopic, Phenotypic and Genetic Characteristics of Adult Patients With Melanoma Diagnosis <40 Years Age. A Prospective, Monocentric Observational Study
Brief Title: Characteristics of Adult Patients With Melanoma Diagnosis <40 Years Age.
Acronym: MELA_2025
Status: Recruiting | Type: Observational
Sponsor: Ente Ospedaliero Ospedali Galliera (Other)
Responsible Party: Principal Investigator, Sanja Javor, Medical doctor, Ente Ospedaliero Ospedali Galliera
Other Study IDs: Melanoma_2025
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Melanoma of Skin
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ARM 1: Patients with melanoma diagnosis aged between 18 and 39 years.

SUMMARY:
The primary objective of the study is to analyse a local cohort of patients aged 18-39 years with melanoma diagnosis in order to determine the prevalence of the disease in this age group.

Secondary objectives are the following:

* To identify risk factors associated with melanoma in young people.
* To characterise the phenotype and dermoscopic features of melanoma in patients aged 18-39 years.
* To analyse the relationship between the clinical and histopathological features of melanoma in young people.
* To identify the mutational status of B-RAF in the sample of patients analysed.

ELIGIBILITY:
Inclusion Criteria:

1. written informed consent
2. age > 18 years and < 40 years
3. diagnosis of cutaneous melanoma even non-primary

Exclusion Criteria:

-

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Since there are no epidemiological data about the prevalence of melanoma in subjects aged 18-39 years, there are very few data available on risk factors in this age group and the impact of the disease.
  The present study, therefore, will enroll about 25 patients who will attend the Dermatology Unit and who have a histological diagnosis of cutaneous melanoma in a period of 24 months of observation.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Melanoma prevalence | 3 years
  Estimated prevalence of melanoma in a cohort group of patients aged 18 - 39 years

SECONDARY OUTCOMES:
Risk factor | 3 years
  Identification of risk factors associated with melanoma in young people.
Melanoma phenotype | 3 years
  Description of the main phenotypic of melanoma in this age group.
Histopathological feature | 3 years
  Evaluation of the likely association between clinical and histopathological features of melanoma in young people.
Mutational status | 3 years
  Identification of the presence of B-RAF mutations
Dermoscopy of melanoma | 3 years
  Description of the main dermoscopic characteristics of melanoma in this age group.

CONTACTS AND LOCATIONS:
Overall Officials: Sanja Javor, Principal Investigator — Ente Ospedaliero Ospedali Galliera
Locations (1):
- E.O. Ospedali Galliera, Genoa, Liguria, Italy

IPD SHARING:
Plan to Share IPD: No